CLINICAL TRIAL: NCT01806818
Title: A Phase 2, Randomized, Double-blind, Parallel, Placebo-controlled, Multi-center Study to Compare Efficacy and Safety Between Eperisone a BID and a TID Regimen in Acute Low Back Pain Patients
Brief Title: Comparing Efficacy and Safety Between Eperisone a BID and a TID Regimen in Acute Low Back Pain Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HM-EPAC-201
Record Dates: First submitted 2013-03-06; First posted 2013-03-07 (Estimated); Last update posted 2013-08-23 (Estimated); Status verified 2013-08

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Eperisone 50mg BID (Experimental): Administrate Eperisone 50mg tablet after the breakfast and dinner, and pacebo tablet after the lunch for 7 days
  Interventions: Drug: Epirisone 50mg or placebo TID
- Epirisone 50mg TID (Experimental)
  Interventions: Drug: Epirisone 50mg or placebo TID
- Placebo comparator (Placebo Comparator)
  Interventions: Drug: Epirisone 50mg or placebo TID

INTERVENTIONS:
Drug: Epirisone 50mg or placebo TID — 3 times a day after meals for 1 week

SUMMARY:
Multi-center Study to Compare Efficacy and Safety between Eperisone a BID and a TID Regimen in Acute Low Back Pain Patients during 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have ability to comprehend the contents of study and before participating in trial and have willingness to sign of informed consent in writing
* 20≤ age ≤60
* A patient has symptom of acute low back pain
* 4≤ VAS

Exclusion Criteria:

* Subjects who cannot prohibit anti-inflammatory drug, painkiller or muscle relaxants during clinical trial
* Chronic rheumatoid arthritis patients
* Patients having a medical history of hypersensitivity to Eperisone Hydrochloride
* Subject having a hereditary problem such as galactose intolerance, Lapp lactase deficiency, or glucose galatose malabsorption
* Participation in other studies before 60 days of first dosing
* Female patients having positive pregnancy test, lactating women,planning pregnancy during clinical trial
* Inadequate subject for the clinical trial by the investigator's decision

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 98 (Actual)
Dates: Start 2013-02; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
VAS improvement of pain at rest, on movement and at night | 7 days

SECONDARY OUTCOMES:
Change of Modified Schober test | 7 days
Change of Lateral Body Bending test | 7 days
Change of EuroQol by patients | 7 days
Change of Oswestry Disability Index | 7 days
Overall pain improvement by investigator | at last visit (D7+2)

CONTACTS AND LOCATIONS:
Overall Officials: Hak-Sun Kim, M.D., Principal Investigator — Gangnam Severance Hospital
Locations (5):
- South Korea (5):
  - Hallym University Sacred Heart Hospital, Anyang
  - CHA Bundang Medical Center, Seoul
  - Kyung Hee University Hospital, Seoul
  - Medical college of Yonsei University, Gangnam Severance Hospital, Seoul
  - Severance Hospital, Seoul